CLINICAL TRIAL: NCT01606488
Title: Effects of Brain Beta Amyloid on Postoperative Cognition and 18F-AV-45-A14: Clinical Evaluation of Florbetapir F 18 (18F-AV-45)
Brief Title: Effects of Brain Beta-Amyloid on Postoperative Cognition
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other); Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20110506; 18F-AV-45-A14 (Other: Avid Radiopharmaceuticals)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Postoperative Cognitive Dysfunction; Postoperative Cognitive Decline; POCD; Alzheimer's disease; Florbetapir F 18 (18F-AV-45)
MeSH Terms: conditions — Postoperative Cognitive Complications; Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical Group (Other): Subjects scheduled to undergo total knee or total hip replacement at the SFVAMC.
  Subjects in this arm of the study will undergo the florbetapir PET scan once prior to their surgery.
  Subjects in this arm of the study will undergo serial neurocognitive assessment, heart rate variability measurement, and blood draws for genetic and inflammatory markers.
  Interventions: Drug: Florbetapir F 18 (18F-AV-45)
- Non-surgical group (Other): Subjects being seen in at the SFVAMC orthopedic clinic for knee or hip pain but are not anticipating surgical intervention.
  Subjects in this arm will not undergo the florbetapir PET scan.
  Subjects in this arm of the study will undergo serial neurocognitive assessment, heart rate variability measurement, and blood draws for genetic and inflammatory markers.
  Interventions: Other: no intervention

INTERVENTIONS:
Drug: Florbetapir F 18 (18F-AV-45) — Single IV bolus injection of 370 MBq (10mCi) florbetapir will be administered approximately 50 minutes prior to a 10 minute PET scan.
  Other Names: Florbetapir; Amyvid 18F-AV-45
  Arms: Surgical Group
Other: no intervention
  Arms: Non-surgical group

SUMMARY:
Postoperative cognitive decline (POCD) affects up to 50% of non-cardiac surgical patients greater than or equal to 65 years of age.

This study will test the hypothesis that preoperative presence of brain beta-amyloid plaques in non-demented subjects increases postoperative cognitive decline (POCD) in elderly subjects scheduled for hip or knee replacement.

The investigators hypothesize that preoperative beta-amyloid plaques will predict postoperative cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for total knee arthroplasty or total hip arthroplasty under general anesthesia (primary arthroplasties and revisions)
* English speaking
* Anticipated stay in the hospital
* Not anticipated to stay intubated postoperatively
* Patients who live with or have regular visits from an individual ("study partner") willing to provide information about the patient's cognitive status
* Willing and able to undergo all testing procedures including neuroimaging and agree to longitudinal follow up
* Adequate visual and auditory acuity to allow neuropsychological testing
* Subjects with Clinical Dementia Rating Scale (CDR) of 0-0.5
* Patients who are not demented
* Subjects sho signed an IRB approved informed consent prior to any study procedures

Exclusion Criteria:

* Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances as indicated by history, which in the opinion of the investigator might pose a potential safety risk to the subject
* Current clinically significant cardiovascular disease.
* History of drug or alcohol abuse within the last year, or prior prolonged history of abuse
* Clinically significant infections disease, including Acquired Immune Deficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV) infection or previous positive test for hepatitis
* History of relevant severe drug allergy or hypersensitivity
* Received an investigational medication under an FDA IND protocol within the last 30 days.
* Current clinically significant unstable medical comorbidities, as indicated by history or physical exam, that pose a potential safety risk to the subject
* Received a radiopharmaceutical for imaging or therapy within the past 24 hours prior to the imaging session for this study
* Severe psychiatric disorders including schizophrenia, bipolar disorders, and major depression as described in DSM-IV within the past year (medical record, GDS score, interview with the patient and study partner)
* Obvious causes for their cognitive impairment (e.g. onset coincides with recent head trauma or stroke)
* Dementia of any cause
* CDR score > 0.5
* Expressed the preference to undergo the procedure under regional anesthesia in form of spinal or epidural anesthesia
* Patients who, in the opinion of the investigator, are otherwise unsuitable for a study of this type

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cognitive Decline | At the time of discharge (or at the latest on the 7th postoperative day)
  Measured using comprehensive neurocognitive test battery

SECONDARY OUTCOMES:
Genetic Polymorphisms | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured by obtaining blood sample
Vagus nerve tone assessment | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using Heart Rate Variability (HRV)
Inflammatory Markers | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured by obtaining blood samples
Perioperative Complications | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Measured using patient medical records
Delirium | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Measured using the Confusion Assessment Method rating scale (CAM) or the CAM-ICU if admitted to the intensive care unit
Coma Assessment | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Measured using the Richmond Agitation Sedation Scale (RASS)
Hospital Length of Stay | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Measured using patient medical records
Postoperative Complications | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using patient medical records
Change in Cognition | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using comprehensive neurocognitive test battery
Quality of Life | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured by assessing functional status using the Functional Activities Questionnaire and depression using the Geriatric Depression Scale
Mortality | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using patient medical records
Pain intensity | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the Numerical Rating Scale
Pain unpleasantness | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the Numerical Rating Scale
Post-traumatic Stress Disorder symptomatology | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the PTSD Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Marek Brzezinski, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No